CLINICAL TRIAL: NCT00983047
Title: Phase II Study of Nimotuzumab Plus Docetaxel in Chemotherapy-refractory/Resistant Patients With Advanced Non-small-cell Lung Cancer
Brief Title: Nimotuzumab Plus Docetaxel in Chemotherapy-Refractory/Resistant Patients With Advanced Non-Small-Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor decide to terminate
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT-IST-NSCLC-010
Record Dates: First submitted 2009-09-21; First posted 2009-09-23 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Advanced Non-Small Cell Lung Cancer
Keywords: Nimotuzumab; NSCLC; Docetaxel
MeSH Terms: interventions — nimotuzumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel (Active Comparator): The chemotherapy treatment:Docetaxel was administered every 3 weeks 75mg/m2, efficacy will be evaluated after two cycles,the chemotherapy will be administered continually 2 cycles if the response is CR\PR\SD. No more than 4 cycles chemotherapy was given.
  Interventions: Drug: Nimotuzumab and Docetaxel
- Nimotuzumab and Docetaxel (Experimental): The chemotherapy treatment:Docetaxel was administered every 3 weeks 75mg/m2,efficacy will be evaluated after two cycles,the chemotherapy will be administered continually 2 cycles if the response is CR\PR\SD.No more than 4 cycles chemotherapy was given.
  Nimotuzumab treatment:Dose of 200mg intravenous infusion per week was continued after the end of chemotherapy until disease progression or unacceptable toxic.
  Interventions: Drug: Nimotuzumab and Docetaxel

INTERVENTIONS:
Drug: Nimotuzumab and Docetaxel — The chemotherapy treatment:Docetaxel was administered every 3 weeks 75 mg/m2, efficacy will be evaluated after two cycles,the chemotherapy will be administered continually 2 cycles if the response is CR\PR\SD. No more than 4 cycles chemotherapy was given.
  Nimotuzumab treatment: Dose of 200 mg intravenous infusion per week was continued after the end of chemotherapy until disease progression or unacceptable toxicity.
  Other Names: Nimotuzumab

SUMMARY:
Nimotuzumab is a humanized monoclonal anti-body targeting the epidermal growth factor receptor (EGFR). Clinical trials are ongoing globally to evaluate nimotuzumab in different indications. Nimotuzumab has demonstrated a unique clinical profile, where anti-tumor activity was observed in absence of severe skin, renal, gastrointestinal mucosa toxicities commonly associated with EGFR-targeting antibodies. Nimotuzumab has been granted approval for use in squamous cell carcinoma of head and neck (SCCHN), glioma and nasopharyngeal cancer in many countries. The investigators compared docetaxel plus nimotuzumab with docetaxel alone in chemotherapy-refractory/resistant patients with advanced EGFR-positive non-small-cell lung cancer to assess the efficacy and safety.

DETAILED DESCRIPTION:
Nimotuzumab and Docetaxel will be administered to the patient until disease progression or unacceptable toxicity had occurred.Docetaxel was administered every 3 weeks 75mg/m2; Nimotuzumab treatment at 200mg per week,at least 12 weeks.The patients'hematology and biochemistry examination will be monitored weekly, a physical exam and assessment of the tumor will be performed and every 6 weeks. The patients will be followed up every 3 months to evaluate the survival.

ELIGIBILITY:
Inclusion Criteria:

1. Histological/cytological confirmed Non-small cell lung cancer
2. EGFR expression is positive (Immunohistochemistry)
3. Locally advanced or advanced NSCLC patients(Stage IIIb \ IV)
4. Patients must have had progressive disease after only one prior chemotherapy regimen.This regimen must have been platinum-based.(For the patients who received new adjuvant chemotherapy or adjuvant chemotherapy, only disease free survival within 9 months will be eligible to enrollment).
5. The last dose of chemotherapy must be finished at least 3 weeks before the study, the acute toxicity of chemotherapy must be recovery.
6. The patients previously received radiotherapy could be recruited. (bone marrow influenced by radiotherapy should be less than 25% of the total quantity of general bone marrow ,and the patients didn't receive the whole pelvis radiation, last radiotherapy must be finished at least 4 weeks before the enrollment. )
7. Patients with at least one tumor lesion that can accurately be measured by magnetic resonance imaging, or computed tomography in at least one dimension with longest diameter to be recorded as ≥ 20 mm using conventional techniques or ≥ 10 mm with spiral CT.
8. ECOG performance status 0-2.
9. Life expectancy ≥ 12 weeks.
10. Adequate organic function must be according with the following:

    * Barrow: Absolute neutrophil count ≥ 1.5×109/L, platelet count ≥ 100×109/L, Haemoglobin ≥ 90g/L;
    * Liver function: BIL ≤ 1.5 x ULN, ALP, AST and ALT≤ 3x ULN or ≤ 5 ULN (Liver metastasis);
    * Renal function: Ccr ≥ 45ml/min;
11. No history of clinically significant or uncontrolled cardiac disease, normal electrocardiogram(ECG).
12. Use of an effective contraceptive method for patients of both genders during study and after the end of 3 months, female subjects must be non breast feeding period and serum or urine pregnancy test should be negative.
13. Signed informed consent and submit to the organization of research

Exclusion Criteria:

1. Brain metastasis and with symptom
2. Previously treatment regimen including:Docetaxel, anti EGFR monoclonal antibody,anti-angiogenesis targeted medicine,small molecule tyrosine kinase inhibitor(TKIs)
3. Receiving other anti-cancer medicine treatment during the study
4. Uncontrolled pleural effusion、seroperitoneum、pericardial effusion
5. Serious illness or other malignancies diagnosed within the past five years.
6. Patients with any serious active infection
7. The second primary malignant tumor
8. Serious accompanying disease would influenced the study (such as cardiac disease,Diabetes mellitus etc)
9. Contraindication of hormone therapy
10. Previous definable peripheral neuropathy and with symptom
11. Do not sign informed consent form

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Median Survival Time | 12 months

SECONDARY OUTCOMES:
Disease control rate | 12 months
Time to progression | 12 months
Safety of the Nimotuzumab and docetaxel (NCI CTC3.0) | 12 months
Quality of life before and after the treatment (QLQ-C30) | 12 months
Analysis EGFR expression, EGFR mutation and amplification, K-ras mutation in the tumor tissues | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University School of Oncology, Beijing Institute for Cancer Research, Beijing Cancer Hospital, Beijing, China